CLINICAL TRIAL: NCT04293445
Title: Phenotyping Asthma Exacerbations: A Longitudinal Cohort Study 2
Brief Title: Asthma: Phenotyping Exacerbations 2
Acronym: APEX 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 19055
Record Dates: First submitted 2019-11-26; First posted 2020-03-03 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: ASTHMA
Keywords: asthma exacerbations
MeSH Terms: conditions — Asthma | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: spirometry, FOT, Induced sputum, bloods, nasal brushes, nasal lavage, skin prick, throat swab — At the point of baseline visit, exacerbation and annual visit, the above tests will be performed to allow comparison of a participants profile before and during an exacerbation

SUMMARY:
The main outcomes of this study are to establish a cohort of well-phenotyped asthma patients with a recent history of an exacerbation. We aim to describe exacerbation profiles (phenotypes) of the cohort in terms of inflammatory/biomarker profile and bacterial/viral infection status and to compare these with exacerbation events in the sister APEX cohort.

DETAILED DESCRIPTION:
A single centre, observational, longitudinal cohort study. The study will consist of one group of approximately 100 patients with clinician diagnosed asthma, who have had at least one exacerbation in the past 5 years before informed consent. They will be identified from secondary care, primary care and the Nottingham Respiratory Research Database (NRRD).

After the Baseline visit, each subject will be followed for the duration of their participation in the study. Participants will be asked to contact the research team if they perceive that their asthma symptoms are worsening to the extent that they would usually seek help from a healthcare professional. They will then be invited to attend the Assessment Visit and potential Exacerbation Visit. Participants who complete this visit will then continue in the study, as we are interested in comparing subsequent events in the same individuals, to establish exacerbation stability and consistency.

All participants, whether they have attended an Assessment visit or not, will be invited to attend for an Annual visit. The research team will also contact participants at 3 monthly intervals, with their permission, to discuss the study and provide updates.

ELIGIBILITY:
INCLUSION

* Clinician diagnosed asthma.
* Male or female aged ≥ 18 and ≤ 85 years of age.
* One asthma exacerbation requiring additional treatment in 5 years prior to informed consent. This is defined as either: 3 or more consecutive day's treatment with oral corticosteroids; for participants not on maintenance steroids, OR at least a doubling of treatment with oral corticosteroids for 3 or more consecutive days, from a stable dose, for participants on maintenance therapy with oral corticosteroids. These can be patient-reported.
* On British Thoracic Society (BTS) step 1-5 treatment
* Current smokers can be included, provided there is good evidence of underlying asthma (for example, a life-long history of asthma, > 12% FEV1 reversibility or sputum or blood eosinophilia).
* Able (in the Investigator's opinion) and willing to comply, with all clinical investigation requirements.
* Non-English speaking participants should be proficient in their understanding of the English language, in order to be able to fully participate in the study.

EXCLUSION:

* Exacerbation in the 4 weeks prior to the Baseline visit. The use of biologic therapy, including Omalizumab, Mepolizumab or Benralizumab, at any time during the 3 months.
* prior to informed consent. Participants who commence biologic therapy during the course of the study will be withdrawn.
* A history more in keeping with smoking-related Chronic Obstructive Pulmonary Disease (COPD)
* Other clinically significant respiratory diseases.
* Use of regular high dose maintenance systemic corticosteroids (for example, a dose of > 10mgs of Prednisolone daily)
* Any other clinically significant medical disease or uncontrolled concomitant disease, that is likely, in the opinion of the investigator, to impact on the ability to participate in the study or the study results.
* Pregnant women, lactating women or women who are planning to become pregnant.
* Participants with uncontrolled hypertension. Participation in a study involving an investigational medicinal product at any time during the 3 months prior to informed consent.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A population of asthmatics who have had an exacerbation in the 60 months prior to the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of study participants with an eosinophilic and non eosinophhilic phenotype | 3 years
  Percentage of study participants with an eosinophilic and non eosinophhilic phenotype

SECONDARY OUTCOMES:
The proportion of exacerbations associated with confrimed viral and bacterial infection | 3 years
  The prercentage of participants within the cohort with at least one exacerbation associated with confirmed viral and bacterial infection by the end of the study
Asthma control questionnaire | 3 years
  ACQ score at baseline and then at exacerbation and annual visits. 0 is total control and 6 is severely uncontrolled
Medication Adherence Rating Scale (MARS) | 3 years
  MARS at baseline and then at exacerbation and annual visits. 5 Questions scored 1-5. 1 being the best and 5 being the worst.
Measuring Lung function and inflammation | 3 years
  Measure Forced Oscialltion Technique (FOT) and Spirometry and Fractional Echaled Nitric Oxide (FENO) at baseline and then at exacerbation and annual visits.
Blood profile | 3 years
  Measure FBC CRP IgE at baseline. During an exacerbation and Annual visit FBC CRP will be measured. Additional bloods will be taken at each visit for future research
Nasal lavage fluid and throat swab | 3 years
  Nasal lavage will be performed along side a throat swab to identify any virsuses at baseline, exacerbation and annual visits.
Skin Prick testing | 3 years.
  Skin prick tests will be performed on all patients at baseline to assess if they are sensitive to common allergens and would be suggestive of atopy
Induced sputum | 3 years
  Induced sputum will be attempted on all patients at baseline exacerbation and on annual visits to assess sputum cell counts at each of the specific points.
Nasal brushes | 3 years
  Nasal brush samples will be obtained to identify viral genetics at baseline, exacerbation and annual visits

CONTACTS AND LOCATIONS:
Overall Officials: Tim Professor Harrison, MBBS, BSc, FRCP, MD, MSc, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham respriatory research unit, Nottingham, Nottinghamshire, United Kingdom